CLINICAL TRIAL: NCT04020302
Title: The Effect of a Self-Monitoring Shopping Intervention for Adults With Intellectual Disability Secondary to Down Syndrome
Brief Title: Self-Monitoring Shopping Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Sharon Gutman, Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS5202
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2019-10

CONDITIONS: Intellectual Disability; Down Syndrome
Keywords: Shopping; Activities of Daily Living
MeSH Terms: conditions — Intellectual Disability; Down Syndrome; Typhus, Endemic Flea-Borne

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shopping group (Experimental): Participants will receive an 8-week intervention which will include weekly sessions that are delivered in an alternating group-individual format. Sessions will provide participants the opportunity to practice and apply self-monitoring techniques across a variety of shopping tasks and settings to promote generalization and transfer of learning (Phase B).
  Interventions: Behavioral: Self-monitoring shopping intervention

INTERVENTIONS:
Behavioral: Self-monitoring shopping intervention — Intervention will occur once per week for a duration of 8 weeks. The intervention format will alternate between individual and group sessions, so that the first week of intervention will be provided in a group format, the second week will be provided in an individual format, and so forth. Sessions will be 90 minutes in duration. Data will be collected during individual sessions, which will occur every other week. During individual sessions, each participant will meet at the facility for the first 15 minutes, will travel to a local grocery store for 45 minutes, and then reconvene at the facility for the final 30 minutes. Group sessions will follow the same structure; however, all ten participants will be present. Each of the 8 sessions will consist of the following: awareness training; facilitation of strategy generation; facilitation of error detection; reinforcement of self-monitoring techniques; and opportunity for participants to practice self-monitoring techniques.

SUMMARY:
The purpose of this study is to examine the effectiveness of a self-monitoring intervention to improve shopping performance in adults with intellectual disability (ID) secondary to Down syndrome (DS). The research question asks, can an 8-week self-monitoring intervention, provided in a community-based setting, increase observable shopping skills in adults with ID secondary to DS?

DETAILED DESCRIPTION:
Adults with intellectual disability secondary to Down syndrome often have difficulty performing complex activities of daily living, such as shopping. These difficulties may, in part, be influenced by deficits in metacognitive abilities, which include self-monitoring of one's performance. There is evidence that interventions which target self-monitoring skills can improve functional performance in adults and adolescents with traumatic brain injury.

Functional magnetic resonance imaging (fMRI) studies on adults with Down syndrome have demonstrated impairments in metacognitive abilities, resulting from significant volume reduction in the frontal lobes and anterior cingulate cortex. These deficits likely contribute to the difficulties experienced by this population when performing instrumental activities of daily living (IADL), such as shopping. Although metacognitive-focused interventions that address self-monitoring skills have been used to improve functional performance in adults and adolescents with traumatic brain injury, these techniques have not yet been used to improve IADL performance in adults with intellectual disability secondary to Down syndrome.

This 16-week study is a single-subject ABA design across ten participants to determine the effectiveness of a self-monitoring intervention on shopping performance in adults with intellectual disability secondary to Down syndrome. The intervention will span 8 weeks and will include weekly sessions that are delivered in an alternating group-individual format. Sessions will provide participants the opportunity to practice and apply self-monitoring techniques across a variety of shopping tasks and settings to promote generalization and transfer of learning. This study has the potential to provide preliminary information on the effectiveness of a self-monitoring intervention, provided in community-based settings, to increase observable shopping skills in adults with intellectual disability secondary to Down syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults with intellectual disability secondary to Down Syndrome
* Members of a community center called GiGi's Playhouse Hillsborough

Exclusion Criteria:

* Severe behavioral disorder that would prevent cooperation with study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with change in level of assistance post intervention | Baseline, up to 8 weeks
  Shopping Skills Recording Sheet will be used to record the level of assistance (5-point ordinal scale) required by participants to demonstrate targeted shopping skills observed in the community. Completion of the instrument requires 25 minutes. There are five levels:
  1. Independent (I) Client performs the task completely without cueing or assistance
  2. Indirect cueing (IC) Therapist provides general information regarding performance, without explicitly stating what is to be done
  3. Direct cueing (DC) Therapist provides specific instructions or feedback about performance
  4. Partial assistance (PA) Client performs part, but not all of the task
  5. Full assistance (FA) Therapist completes the task for the client in its entirety

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gutman, PhD, Principal Investigator — Professor of Rehabilitation and Regenerative Medicine
Locations (1):
- GiGi's Playhouse Hillsborough, Hillsborough, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No